CLINICAL TRIAL: NCT04996108
Title: An Observational Study to Investigate the Auto-inflammatory Basis of Recurrent Pericarditis
Brief Title: Pericarditis: Auto-Inflammation in Recurrent Disease
Acronym: PAIReD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 286959
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Idiopathic Recurrent Pericarditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Participants with recurrent pericarditis (RP): Patients aged 16 or over with (1) RP, diagnosed by a clinician, meeting the European Society of Cardiology (ESC) diagnostic criteria, and (2) where the aetiology of the RP is defined as idiopathic (i.e. there is no other aetiology identified, such as infective, malignant, post cardiac injury, as part of an autoimmune condition, as part of another known auto-inflammatory disease).
- Participants with systemic auto-inflammatory diseases (disease controls): Patients aged 16 or over with a systemic auto-inflammatory disease, diagnosed by a trained specialist.
- Healthy volunteers (healthy controls): Sex, ethnicity and aged matched healthy individuals who do not have a personal history of pericarditis or systemic auto-inflammatory disease.
- Relatives of individuals with recurrent pericarditis (familial controls): First degree relatives of participants meeting the criteria for, and included in the study as, RP cases, who are aged 16 or over.

SUMMARY:
Pericarditis is swelling of the sac that surrounds the heart, the pericardium, causing chest pain. For most patients, the condition improves with simple anti-inflammatory medications like colchicine and ibuprofen. However, in 20-30% of patients the condition comes back. Diagnosis of recurrent pericarditis is frequently missed or delayed, and many patients require prolonged courses of corticosteroids to control their disease. Together these factors damage the quality of life of patients with recurrent pericarditis. Currently there is limited understanding of why pericarditis comes back in some patients, and how best to treat it when it does.

PAIReD (Pericarditis: Auto-Inflammation in Recurrent Disease) is an observational research study funded by the British Heart Foundation that will investigate the role inflammation plays in recurrent pericarditis. Patients with recurrent pericarditis and other auto-inflammatory diseases will be recruited from the specialist fever clinic at the Royal Free Hospital, where they will be asked to donate blood up to six times over a three year period. Healthy participants will be recruited at the Royal Free Hospital or Guy's Hospital. Relatives of participants with recurrent pericarditis will be recruited at the Royal Free Hospital. They latter two groups will attend one appointment where blood or saliva samples will be taken. A subset of participants will also provide fingerstick blood samples and questionnaires from home, for up to one year.

Clinical data will be collected prospectively and by retrospective case note review. Blood from participants will be analysed to look at how the immune cells of patients with recurrent pericarditis function during the course of their disease, and to look for genetic changes in patients with recurrent pericarditis that might contribute to their condition. Together this knowledge has to potential to help clinicians diagnose and monitor patients with recurrent pericarditis more accurately, and researchers to design more effective treatments.

ELIGIBILITY:
Inclusion Criteria:

Recurrent pericarditis (RP) cases:

1. Patients with RP, diagnosed by a clinician, meeting the European Society of Cardiology (ESC) diagnostic criteria.
2. Where the aetiology of the RP is defined as idiopathic (i.e. there is no other aetiology identified, such as infective, malignant, post cardiac injury, as part of an autoimmune condition, as part of another known auto-inflammatory disease).

Relatives of RP cases:

First degree relatives of participants meeting the criteria for, and included in the study as, RP cases.

Disease Controls:

Patients with a systemic auto-inflammatory disease, diagnosed by a trained specialist.

Healthy Controls:

Sex, ethnicity and aged matched healthy individuals who do not have a personal history of pericarditis or systemic auto-inflammatory disease.

Exclusion Criteria:

1. Individuals under 12 years of age
2. Adults who are unable to give written informed consent
3. Individuals who have received a blood transfusion within 4 weeks

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population for cases comprises patients under the care of the recruiting sites with a diagnosis of RP.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2021-07-29 (Actual); Primary Completion 2024-06-13 (Estimated); Study Completion 2024-06-13 (Estimated)

PRIMARY OUTCOMES:
Immune cell phenotype | Three years
  Exploratory analysis of the proportion, maturity and activation state of different immune cell populations in the peripheral blood, comparing cases and controls and correlated to disease activity in cases
Immune cell gene expression | Three years
  Exploratory analysis of the transcriptome in immune cells in cases compared to controls, and correlated to disease activity in cases.

SECONDARY OUTCOMES:
Genotype | Three years
  Candidate gene analysis and whole exome sequencing of cases and familial controls.
Clinical phenotype | Three years
  Characterisation of clinical course of cohort of RP patients, gathering data on disease activity and quality of life prospectively over three years

CONTACTS AND LOCATIONS:
Overall Officials: Claire J Peet, BMBCh MRCP, Principal Investigator — Clinical research fellow
Locations (2):
- United Kingdom (2):
  - Royal Free Hospital NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London